CLINICAL TRIAL: NCT02594761
Title: Pharmacokinetic Study Comparing Hercules, EU-approved Herceptin® and US-Licensed Herceptin® Administered as a Single Intravenous Infusion to Healthy Male Volunteers
Brief Title: Phase 1 Study of Trastuzumab Administered as a Single Intravenous Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Myl-Her 1002
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — hercules receptor kinase 2, Arabidopsis; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Hercules: 8 mg/kg i.v. infusion over 90 minutes
  Interventions: Biological: Hercules
- Treatment B (Active Comparator): Herceptin EU: 8 mg/kg i.v. infusion over 90 minutes
  Interventions: Biological: Herceptin EU
- Treatment C (Active Comparator): Herceptin US: 8 mg/kg i.v. infusion over 90 minutes
  Interventions: Biological: Herceptin US

INTERVENTIONS:
Biological: Hercules — Powder Concentrate for Intravenous Infusion, 150 mg/vial
  Other Names: Trastuzumab
  Arms: Treatment A
Biological: Herceptin EU — Powder for Concentrate for Solution for Infusion, 150 mg/vial
  Other Names: Trastuzumab
  Arms: Treatment B
Biological: Herceptin US — Intravenous Infusion, 440 mg/vial
  Other Names: Trastuzumab
  Arms: Treatment C

SUMMARY:
The primary objective of this study was to demonstrate pharmacokinetic similarity of Mylan trastuzumab (Hercules) versus EU-approved Herceptin® and US-licensed Herceptin® and pharmacokinetic similarity of EU-approved Herceptin® versus US-licensed Herceptin® after 8 mg/kg as single dose administered as intravenous infusion over 90 minutes in healthy male subjects based on the equivalence criterion that AUC0-∞, AUC0-last, and Cmax least square mean ratios are bounded within the 90% confidence intervals, 80.00% - 125.00%. Three similarity assessments were performed, 1) Hercules vs. EU-approved Herceptin®, 2) Hercules vs. US-licensed Herceptin® and 3) EU-approved Herceptin® vs. US-licensed Herceptin®. Secondary objectives included further pharmacokinetic assessment of similarity of Hercules, EU-approved Herceptin® and US-licensed Herceptin® λz, tmax and t1/2 along with assessment of safety (including immunogenicity) and local tolerance.

DETAILED DESCRIPTION:
All subjects checked into the clinical facility on the day prior to dosing. On study day 1, each subject received either a single i.v. infusion of 8 mg/kg BW in 250 mL normal saline over a 90 minute period of Mylan trastuzumab (Hercules), EU-approved Herceptin®, or US-licensed Herceptin®. Dosing occurred following an overnight fast of at least 8 hours. On the day of dosing, subjects fasted for the first 3 hours after the start of the infusion then received standard meals approximately 3, 6 and 9 hours post-dose. In each study period, blood samples were collected just immediately prior to dose administration (0 hour) and at 45 and 90 minutes (just prior to end of infusion). Blood samples were collected post-dose at 3, 6, 9, 24 and 48 hours, relative to the start of infusion. The subjects were allowed to leave the clinical facility after the 48-hour blood sample collection. Subjects returned to the clinical facility for the scheduled blood sample collections post-dose on Day 5, 8, 11, 15, 22, 29, 43, 57, and 71. Serum samples were stored at -80°C ± 15°C until shipment for analysis. Blood samples for anti-drug antibodies (ADA) were collected prior to dosing on Day 1 and on Day 71. Blood samples for C-reactive protein (CRP) were obtained at Screening, prior to dosing and at 3, 24 and 48 hours post-dose and on Day 8 and 71. Blood samples for analysis of immunoglobulins were collected prior to dosing on Day 1 and on Day 8 and 71.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects, age 18 to 55 years old
* able to understand procedures, agree to participate and willing to give informed consent

Exclusion Criteria:

* history of any significant disease
* use of any medication 7 days prior to start of study
* participation in a clinical trial within 30 days of start of study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 71 days
  The primary pharmacokinetic variables for assessment of bioequivalence are dose-normalized Cmax based on the equivalence criterion that Cmax least square mean ratios are bounded within the 90% confidence intervals, 80.00% - 125.00%.
Area Under the Plasma Concentration Versus Time Curve (AUC) - Time 0 to Last Blood Draw (AUC0-last) | 71 days
  The primary pharmacokinetic variables for assessment of bioequivalence are dose-normalized AUC0-last based on the equivalence criterion that AUC0-last least square mean ratios are bounded within the 90% confidence intervals, 80.00% - 125.00%.
Area Under the Plasma Concentration Versus Time Curve (AUC) - Time 0 to Infinity AUC0-∞) | 71 days
  The primary pharmacokinetic variables for assessment of bioequivalence are dose-normalized AUC0-∞, based on the equivalence criterion that AUC0-∞ least square mean ratios are bounded within the 90% confidence intervals, 80.00% - 125.00%.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) | 71 days
Local Infusion Tolerance | 71 days
Immunogenicity | 71 days
Measurement of C-reactive Protein | 71 days
Monitoring of Heart Function (ECG and Echocardiography) | 71 days

CONTACTS AND LOCATIONS:
Overall Officials: Apinya Vutikullird, D.O., Principal Investigator — WCCT Global

REFERENCES:
- [Derived] Waller CF, Vutikullird A, Lawrence TE, Shaw A, Liu MS, Baczkowski M, Sharma R, Barve A, Goyal P, Donnelly C, Sengupta N, Pennella EJ. A pharmacokinetics phase 1 bioequivalence study of the trastuzumab biosimilar MYL-1401O vs. EU-trastuzumab and US-trastuzumab. Br J Clin Pharmacol. 2018 Oct;84(10):2336-2343. doi: 10.1111/bcp.13689. Epub 2018 Jul 31. PMID 29926514